CLINICAL TRIAL: NCT04517760
Title: Evaluating an HIV Risk Screening Tool for Use in a Population of Orphans and Other Vulnerable Children in Tanzania
Brief Title: Evaluating an HIV Risk Screening Tool for Orphans and Vulnerable Children in Tanzania
Status: Completed | Type: Observational
Sponsor: Elizabeth Glaser Pediatric AIDS Foundation (Other)
Collaborators: Tanzania Ministry of Health, Community Development, Gender, Elderly and Children (Unknown); PACT International (Unknown)
Responsible Party: Sponsor
Other Study IDs: EG0216
Record Dates: First submitted 2020-08-12; First posted 2020-08-18 (Actual); Last update posted 2020-08-18 (Actual); Status verified 2020-08

CONDITIONS: Pediatric HIV Infection
Keywords: HIV Screen tool; orphans and vulnerable children; Tanzania

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of the research was to evaluate the performance of items within the Kizazi Kipya (K2) Orphan and Vulnerable Children (OVC) HIV risk screening tool in identifying HIV-positive children, to optimize an HIV screening tool for OVC and children and adolescents in facility settings and to assess the feasibility and acceptability of home-based HIV risk screening and testing.

DETAILED DESCRIPTION:
Under the ongoing community-based Kizazi Kipya (K2) OVC project, program staff currently administer a 13-item HIV risk screening tool to all K2 program beneficiaries, and refers those who screen positive to facility-based HIV testing. A subset of this 13-item tool is a module of four items that had previously been used as a standalone four-question screening tool in facilities in Zimbabwe.

The primary objectives of this study are as follows.

1. To evaluate the performance of a lay cadre-administered four-item subset of the K2 HIV risk screening tool that matches the Zimbabwe evidence-based tool in predicting the HIV status of vulnerable children/adolescents represented by two populations: (a) K2 OVC beneficiaries and (b) children/adolescents attending health facilities.
2. To identify additional items in the K2 HIV risk screening tool that could be added to the four-question subset to improve the tool's performance.
3. To assess fidelity to the administration of the OVC HIV screening tool items through structured observations of community case workers in the K2 program.
4. To assess the acceptability of OVC HIV risk screening and testing implemented in the community among OVC beneficiaries in the K2 program.
5. To assess the acceptability and feasibility of integrating the OVC HIV screening tool with HIV testing among OVC community case workers in the K2 program.

ELIGIBILITY:
Children and adolescents and their caregivers:

Inclusion Criteria:

* Living in a household deemed to be at elevated HIV risk based on previously identified risk criteria
* Attending a study health facility in two regions of Tanzania
* Age 2-19 years

Exclusion Criteria:

* Previously tested HIV-positive
* History of antiretroviral treatment (ART)
* Unable or unwilling to be consented
* Age 5-19 years old, tested negative in past 6 months, and having no reported exposure to HIV through sexual contact (consensual, abuse) or through blood transfusion/needle injury.

Community care workers:

Inclusion criteria:

* conducting HIV risk screening in OVC households as part of their role in the Kizazi Kipya project in the subset of study districts where structured observations and focus group discussions were conducted

Exclusion criteria:

* unwilling to consent to the study

Ages: 2 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children and adolescents (and their caregivers as applicable) participating in an orphans and vulnerable children (OVC) program or presenting for services at a study facility. Community care workers (CCWs) who have been conducting HIV risk screening in OVC households as part of their role in the OVC program.
Sampling Method: Non-Probability Sample
Enrollment: 21080 (Actual)
Dates: Start 2018-02-22 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Sensitivity of HIV risk screening tool | Within four weeks
  Children/adolescents testing HIV positive on the tool who are truly HIV positive
Specificity of HIV risk screening tool | Within four weeks
  Children/adolescents testing HIV negative on the tool who are truly HIV negative
Positive predictive value | Within four weeks
  Proportion of children/adolescents testing positive on the tool who actually have HIV
Negative predictive value | Within four weeks
  Proportion of children/adolescents testing negative on the tool who do not actually have HIV
Acceptability of HIV risk screening tool | Within six weeks
  Examining the extent of reception of the screening tool by the OVC caregivers and the community case workers using a semi-structured questionnaire
Feasibility of HIV risk screening tool | Within six weeks
  Exploring the practicality of use of HIV risk screening tool through focus group discussions with community case workers

CONTACTS AND LOCATIONS:
Overall Officials: Gretchen Antelman, PhD, Principal Investigator — E. Glaser Pediatric AIDS Found
Locations (1):
- Elizabeth Glaser Pediatric AIDS Foundation, Dar es Salaam, Tanzania

IPD SHARING:
Plan to Share IPD: Yes
The IPD sharing plan will include the final quantitative datasets, tools, data dictionaries and analytic code will be made publicly available through a Dataverse repository.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: End 2020
Access Criteria: Dataverse repository